CLINICAL TRIAL: NCT05623891
Title: Safety Study of 177Lu-Anti-ED-B mAbs SPECT Imaging in Patients With ED-B Positive Solid Tumors
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Affiliated Hospital of Jiangnan University (Other)
Responsible Party: Principal Investigator, Chunjing Yu, Director, Affiliated Hospital of Jiangnan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LS2022026
Record Dates: First submitted 2022-11-07; First posted 2022-11-21 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 177Lu-Anti-ED-B mAbs (Experimental): Patients will receive a tracer (5 mg, IV) dose of 177Lu (10 mCi) labeled anti-ED-B mAbs(177Lu-B5-IgG4)
  Interventions: Drug: 177Lu-B5-IgG4

INTERVENTIONS:
Drug: 177Lu-B5-IgG4 — 177Lu-B5-IgG4 injection followed by SPECT scan

SUMMARY:
This is a single arm study to evaluate the safety and biodistribution of 177Lu-labeled anti-ED-B mAbs SPECT imaging in patients with ED-B positive solid tumors.

DETAILED DESCRIPTION:
After being fully informed about the study and potential risks, all patients giving written informed consent will be evaluated to determine eligibility for study entry. Patients will receive an injection of 177Lu-labeled anti-ED-B mAbs and will undergo SPECT/CT scanning to determine uptake of 177Lu-labeled anti-ED-B mAbs in tumor lesions and normal tissues and organs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily signed informed consent, and be able to complete the trial according to the requirement of the scheme;
2. Aged 18-75, male or female;
3. Patients diagnosed with solid tumors confirmed by histopathology ;
4. Patients with biopsy-proven fibronectin ED-B positive;
5. At least one measurable solid lesions has been examined by 18F-FDG PET/CT (RECIST1.1 standard);
6. ECOG score 0~2;
7. ALT, AST shall not exceed 3 times of the normal upper limit; Bun, Cr not exceed 1.5 times of the normal upper limit.
8. Other routine examinations are within the normal range or considered acceptable by the researchers.

Exclusion Criteria:

1. Recovery from major trauma (including surgery) within 4 weeks prior to study treatment;
2. Patients with systemic or locally severe infections, or other serious coexisting diseases;
3. Patients with abnormal immune function or who have recently used immunosuppressive or potentiating agents including various vaccines;
4. Patients with autoimmune diseases, including rheumatoid arthritis;
5. Inadequate control of arrhythmias, including atrial fibrillation;
6. Uncontrolled hypertension;
7. Patients with allergies or allergies to any component of the imaging agent or antibody;
8. Patients who cannot undergo PET/CT imaging scan;
9. Syphilis, HBV, HCV, or HIV positive subjects;
10. Male and female subjects of reproductive age cannot take effective contraceptive measures;
11. Pregnant or lactating women;
12. Patients with a history of mental illness or related conditions;
13. Other subjects considered unsuitable by researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of tissue distribution of 177Lu-Anti-ED-B mAbs(B5-IgG4) | 1 year
  Biodistribution of 177Lu-Anti-ED-B mAbs(B5-IgG4) evaluated by radioactive uptake values (standardized uptake values, SUVs) in various organs during repeated 177Lu-SPECT scans will be reported.
Dosimetry estimates of 177Lu-Anti-ED-B mAbs(B5-IgG4) | 1 year
  Absorbed dose (radioactive uptake) estimates for different organs and tissues calculated with the AUCs and the OLINDA/EXM dosimetry program will be obtained and reported.
Incidence of Treatment-Emergent Adverse Events | 1 year
  Safety will be assessed by evaluation of incidence of adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No